CLINICAL TRIAL: NCT00142311
Title: Clinical, Molecular and Metabolic Comparison Between Early Onset Parkinsonian, With or Without Parkin Mutation: Physiopathological Perspectives
Brief Title: Functional Characterization of Parkin + Patients
Status: Terminated | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Other Study IDs: A02094; 4CC03H-A02094SP; RAF/03003/P011104/PCR02006
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Parkin mutations; Metabolic explorations; Clinics; Genetics
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Parkinson's disease is one of the most frequent neurodegenerative diseases, and for which the mechanisms remains unknown. Since the implication of susceptibility factors is highly suspect, we have recently shown that one monogenic form due to alterations in the Parkin gene was responsible for an important proportion of early onset familial and isolated cases. Nevertheless, it not has been determined yet the relationship between idiopathic Parkinson's disease and secondary Parkinson's disease with a Parkin gene mutation at the clinical, neuropsychological, metabolic and physiopathological levels. For establishing phenotype-genotype correlations, we propose to compare the phenotype of patients carrying a Parkin mutation (parkin " + ", n=25) to those of early onset parkinsonians without a Parkin mutation (Parkin " - ", n = 25), and for some aspects (neuropsychological, behavioural and psychiatric evaluations) to the healthy brothers and sisters of Parkin cases "+"(n = 25). The evaluation will carry on the clinical aspects (quantification of the parkinsonian syndrome and reactivity to levodopa, neuropsychological, behavioural and psychiatric evaluations), molecular (types of abnormalities in the Parkin gene) and metabolic (PET - tomography by positron emission) of the disease.

Parkinson's disease caused by Parkin gene mutations is associated with an important and homogeneous loss of dopaminergic neurons of the substantia nigra pars compacta, which is different from those observed during the idiopathic Parkinson's disease. The corresponding dopaminergic deficit should be associated with an excellent reactivity to levodopa, to a cognitive deficit and to behavioural and/or psychiatric attitudes, in relation with the massive alteration of dopaminergic efferences.

This multidisciplinary approach on Parkin cases will be performed in the centers for of clinical investigations of Grenoble and Paris, with the help of the French Parkinson's Disease Study Group, and two centers for TEP (Lyon and Orsay). This project will allow to a better definition of diagnostic criteria of Parkin " + " cases, which will help for the molecular diagnosis in early onset cases, and will study precisely the clinical, psychiatric and metabolic consequences of a massive and homogeneous dopaminergic denervation, which seems to be different of idiopathic Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

- Age at onset before 45 Presence of at least two of the three cardinal signs: bradykinesia, rigidity with dental wheel, postural tremor Frank response to L-Dopa (> 30 %) Absence of personal history of meningitis-encephalopathy, neuroleptic treatment, absence of pyramidal, cerebellar or oculomotor signs, absence of dysautonomia or dementia that occurred less than 2 years before the onset of the disease Exclusion of Wilson's disease by usual biological tests Normal cerebral MRI

Exclusion Criteria:

- Incapacity of the patient to understand and participate in the protocol

Patients who present a contraindication to the realization of cerebral MRI (pacemaker, cardiac valve, ustensile of neurosurgery or vascular surgery, intraocular tissue) could not be included in the group of patients with PET.

Women in age to procreate could not participate to the study with PET, only if she uses an effective contraception (oestroprogestives or a coil). Furthermore, the dates of PET examinations should be at the beginning of the menstrual cycle. At the first doubt, a dosage of b-HCG will be performed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97
Dates: Start 2003-11; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Brice, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris, University Paris 6
Locations (14):
- France (14):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU, Grenoble
  - Hôpital Roger Salengro, Lille
  - Hôpital Neurologique Pierre Wertheimer, Lyon
  - Hôpital René et Guillaume Laennec, Nantes
  - Hôpital Saint-Antoine, Paris
  - Pitié-Salpêtrière Hospital - Centre of Clinical Investigations, Paris
  - Pitié-Salpêtrière Hospital - Federation of Neurology, Paris
  - Pitié-Salpêtrière Hospital - Service of Psychiatry, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Hôpital Pontchaillou, Rennes
  - Hôpital Civil, Strasbourg
  - Hôpital Purpan, Toulouse

REFERENCES:
- See also: Related Info — http://www.inserm.fr